CLINICAL TRIAL: NCT00608660
Title: Studying of Acupuncture for Bell's Palsy According to Different Stages
Brief Title: Randomized Controlled Trial of Acupuncture to Treat Bell's Palsy According to Different Stages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: LiYing, Acupuncture & Tuina college of chengdu univeristy of TCM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006BAI12B03
Record Dates: First submitted 2008-01-04; First posted 2008-02-06 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Bell's Palsy
Keywords: Peripheral Facial Paralysis; Acupuncture; RCT
MeSH Terms: conditions — Bell Palsy; Facial Paralysis | interventions — Acupuncture Therapy; Moxibustion; Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A (Experimental): staging acupuncture for treating Bell's Palsy
  Interventions: Other: acupuncture
- B (Experimental): staging acupuncture and moxibustion for treating Bell's Palsy
  Interventions: Other: acupuncture and moxibustion
- C (Experimental): staging electroacupuncture for treating Bell's Palsy
  Interventions: Other: electroacupuncture
- D (Experimental): staging acupuncture along Yangming musculature for treating Bell's Palsy
  Interventions: Other: acupuncture along yangming tendons
- E (Experimental): non-staging acupuncture for treating Bell's Palsy
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — staging acupuncture
  Arms: A
Other: acupuncture and moxibustion — staging acupuncture and moxibustion
  Arms: B
Other: electroacupuncture — staging electroacupuncture
  Arms: C
Other: acupuncture along yangming tendons — staging acupuncture along Yangming musculature
  Arms: D
Other: acupuncture — non-staging acupuncture
  Arms: E

SUMMARY:
The purpose of this trial will certify the efficacy of using staging acupuncture and moxibustion to treat Bell's Palsy

DETAILED DESCRIPTION:
The result of this trial (available in 2009) aims to testify the efficacy of using staging acupuncture and moxibustion to treat Bell's Palsy, and to approach a best acupuncture treatment among these five different methods for treating Bell's Palsy

ELIGIBILITY:
Inclusion Criteria:

* patients who meet the diagnosis, stages, location criteria
* the first time to onset the disease
* between 1 and 70 days with the onset time of facial palsy
* on one side of the face paralysis
* between 15 and 70 years old with the onset age of facial palsy
* willing to finish the whole observation period
* with written consent form signed by themselves.

Exclusion Criteria:

* facial palsy caused by other disease, such as infectivity multiple radiculitis, tumor which offend temporal bone, cerebral trauma
* facial palsy combine diabetes, the severe disease of heart vessel, cerebral vessel, liver, kidney, lung, and psychosis
* patient with Hunt's syndrome
* patient with facial spasm
* pregnant women or women in lactation
* patients are participating other clinical research

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
House-Brackmann scale （Global Score） | a week

SECONDARY OUTCOMES:
Classification Score Of Facial Paralysis Degree | a week
Facial Disability Index | a week
WHOQOL-BREF scale | two week
House-Brackmann scale （Regional Score） | a week

CONTACTS AND LOCATIONS:
Overall Officials: Ying Li, Dr., Principal Investigator — Acupuncture&Moxibustion college of chengdu TCM
Locations (1):
- Chengdu university of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhao L, Zhang FW, Li Y, Wu X, Zheng H, Cheng LH, Liang FR. Adverse events associated with acupuncture: three multicentre randomized controlled trials of 1968 cases in China. Trials. 2011 Mar 24;12:87. doi: 10.1186/1745-6215-12-87. PMID 21435214